CLINICAL TRIAL: NCT01464346
Title: A Performance Evaluation of the Enlite Glucose Sensor to Support a Full 144 Hours(6Days) of Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEP247
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
Keywords: diabetes; glucose sensor; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Enlite sensor, Abdomen/Abdomen (Experimental): Subjects wearing 2 Enlite sensors in Abdomen
  Interventions: Device: Enlite Sensor
- Enlite sensor, Abdomen/Buttock (Experimental): Subjects wearing 2 Enlite sensors in Abdomen/Buttock
  Interventions: Device: Enlite Sensor
- Enlite sensor, Buttock/Buttock (Experimental): Subjects wearing 2 Enlite sensors in Buttock/Buttock
  Interventions: Device: Enlite Sensor

INTERVENTIONS:
Device: Enlite Sensor — This is the Enlite sensor (all subjects)

SUMMARY:
The purpose of this study is to demonstrate the performance of the Enlite Sensor over an entire calibration and wear period of 146 hours (6 days) when inserted in the abdomen and buttock and used with the Revel 2.0 Pumps in subjects age 18 - 75 years.

DETAILED DESCRIPTION:
The study is a multi-center, prospective single-sample correlational design without controls. Between 4 and 10 investigational sites will be used during this study. All subjects will be assigned to treatment. Each subject will wear the following devices:

1. Enlite Sensors (2) connected to MiniLinks (2)
2. Revel 2.0 Pumps (2)

During the study each subject will be wearing 2 sensors and 2 pumps simultaneously. The pumps will be differentiated by color, and will have different calibration requirements during the in-clinic portions of the study. During the Frequent Sampling Tests:

* GREEN pump will be calibrated 3-4 times spread throughout the day
* RED pump will have the minimum calibration requirements (every 12 hours after the second calibration)

During home use (outside the clinic) BOTH pumps will be calibrated 3-4 times spread throughout the day.

Sensors will be connected to the MiniLink (integrated with the Revel 2.0 Pumps)

Subjects will wear the devices for a 3-day training period, followed by a 6-day study period. During the study period, each subject will undergo three 12-hour Frequent Sampling Tests. During the Frequent Sampling Tests, IV blood samples will be drawn every 5-15 minutes and analyzed using the YSI. The Frequent Sampling Tests will occur during the following hours of sensor wear: hours 2-14, hours 14-26, hours 50-62 hours 62-74, and hours 122-134 hours 134-146 which is representative of a complete calibration and wear period to support the proposed labeling claim of 144 hours of use.

Even though participants were randomly assigned with respect to timing of frequent sample test and sensor insertion locations, data was collected as a whole and there was no intention to analyze the two groups separately. Please note that subjects were randomly assigned to one of 3 different sensor insertion site combinations: abdomen/abdomen, buttock/buttock, and abdomen/buttock

During each Frequent Sampling Test, subjects with an established insulin sensitivity ratio and insulin carbohydrate ratio will undergo a hypoglycemic challenge (glucose lowered to a target of 50-75 mg/dL for ~2 hours, including 30 minutes between 50-60 mg/dL) and a hyperglycemic challenge (glucose raised to a target of 180-400 mg/dL for ~2 hours, including 30 minutes between 350 -400 mg/dL). Subjects will continue with their current diabetes regimen (including glucose monitoring with their own meter when desired) independent of the study devices. The Revel 2.0 Pumps will not be used to infuse insulin or manage the subject's diabetes during this study. The Enlite Glucose sensor will not be used to manage the subject's diabetes during this study. The investigational Study Meter may be used for confirmation of alarms, treatment decisions and calibration of sensor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 - 75 years of age at time of screening
2. A clinical diagnosis of type 1 or 2 diabetes as determined by the

   Investigator, for a minimum of 12 months duration:
   * Criteria for type 1 diabetes:

     * Required: Age of onset < 40 years of age
     * Required: History of insulin use only for management of diabetes
     * Required: history of normal weight or underweight at time of diagnosis.
     * Not required: Initial presentation of diabetic ketoacidosis.
     * Not required: History of diabetic ketoacidosis
     * Not required: Low fasting C-peptide
   * Criteria for type 2 diabetes:

     * Required: Age of onset ~ 40 years of age
     * Required: History of initial oral anti-diabetic use
     * Required: History of being overweight at time of diagnosis.

       * Type 2 insulin requiring is defined by type 2 diabetes subjects taking insulin with or without oral anti-diabetic agent and may also include: incretin mimetic, pramlintide or GLP agonist
       * Type 2 non-insulin requiring is defined by type 2 diabetes subjects who take oral medications and may also include: incretin mimetic, pramlintide or GLP agonist
3. Adequate venous access as assessed by investigator or appropriate staff

Exclusion Criteria:

1. Subject is unable to tolerate tape adhesive in the area of sensor placement.
2. Subject has any unresolved adverse skin condition in the area of sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject has a positive pregnancy screening test
5. Subject is female and plans to become pregnant during the course of the study
6. Subject has had a hypoglycemic seizure within the past 6 months
7. Subject has a history of a seizure disorder
8. Subject has central nervous system or cardiac disorder resulting in syncope
9. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
10. Subjects with hematocrit lower than 36%
11. SUbjects with a history of any cardiac arrhythmia, including atrial arrhythmias
12. Subjects with a history of adrenal insufficiency
13. Subjects with migraines

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lee, MD, Study Director — Medtronic Diabetes
Locations (7):
- United States (7):
  - Profil Institute for Clinical Research, Chula Vista, California
  - AMCR Institue, Escondido, California
  - University of California, San Diego, La Jolla, California
  - Diablo Clinical Research, Walnut Creek, California
  - University of Colorado Denver/Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Oregon Health & Science University, Portland, Oregon
  - Rainier Clinical Research Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enlite Sensor Abdomen/Abdomen: Subjects wearing 2 Enlite sensors in abdomen. Some subjects participated in Frequent Sampling Tests during the first 12 hours of days 1, 3 and 6 while others participated during the last 12 hours of days 1, 3, and 6.
- Enlite Sensor Abdomen/Buttock: Subjects wearing one Enlite sensor in Abdomen and one Enlite sensor in Buttock. Some subjects participated in Frequent Sampling Tests during the first 12 hours of days 1, 3 and 6 while others participated during the last 12 hours of days 1, 3, and 6.
- Enlite Sensor Buttock/Buttock: Subjects wearing 2 Enlite sensors in Buttock. Some subjects participated in Frequent Sampling Tests during the first 12 hours of days 1, 3 and 6 while others participated during the last 12 hours of days 1, 3, and 6.
Period: Overall Study
Arm/Group | Enlite Sensor Abdomen/Abdomen | Enlite Sensor Abdomen/Buttock | Enlite Sensor Buttock/Buttock
Started | 29 | 32 | 29
Completed | 29 | 32 | 28
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects Entering the Study: All Subjects who provided consent, met inclusion/exclusion criteria and worn Enlite sensors
Arm/Group | All Subjects Entering the Study
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 82
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 90

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Agreement (Percent of Sensor Values Within 30% of Reference Value) With Minimum Calibration, Combined Abdomen and Buttock Insertion Sites
Description: Primary endpoint is mean of daily percentage of sensor values within 30% of reference value (within 22.5 mg/dL if YSI <75 mg/dL) with the minimum calibration (every 12 hour), combined abdomen and buttock insertion sites across all participants and all days.
Time Frame: Days 1, 3 and 6 of sensor wear
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Groups:
- All Subjects: This group contains all subjects that enrolled in the study
Arm/Group | All Subjects
Number analyzed (Participants) | 90
percentage of paired readings | 88.01 [85.69 to 90.33]
Statistical Analysis 1: Comparison: All Subjects; Test type: Superiority or Other; p < 0.05, ANCOVA; Mixed effects model was used, with day of sensor wear(1,3 or 6) as covariate. Day was centered to 0 to permit interpretation of the model intercept; Intercept from ANCOVA as agreement rate = 88.01, 95% CI 2-sided [85.69 to 90.33], Standard Error of Mean 1.2

2. Secondary Outcome: Mean Daily Agreement (Percent of Sensor Values Within 30% of Reference Value) With 3-4 Calibrations Per Day, Combined Abdomen and Buttock Insertion
Description: Secondary endpoint is mean of daily percentage of sensor values within 30% of reference value (within 22.5 mg/dL if YSI <75 mg/dL) with 3-4 calibrations per day, combined abdomen and buttock insertion sites across all participants and all days.
Time Frame: Days 1, 3 and 6 of sensor wear
Measure: Mean (95% Confidence Interval); unit: percentage of paired readings
Arm/Group | All Subjects
Number analyzed (Participants) | 90
percentage of paired readings | 90.52 [88.77 to 92.28]
Statistical Analysis 1: Comparison: All Subjects; Test type: Superiority or Other; p < 0.05, ANCOVA; [statistical method as in outcome 1, analysis 1]; Intercept from ANCOVA as agreement rate = 90.52, 95% CI 2-sided [88.77 to 92.28], Standard Error of Mean 0.9

3. Other Pre Specified Outcome: Mean Absolute Relative Difference (MARD) Between Sensor and YSI for Abdomen Insertion Site, With 3-4 Calibrations Throughout the Day
Description: This measure is the Mean Absolute Relative Difference (MARD) between sensor glucose values and and paired YSI plasma glucose values for Abdomen insertion site, with 3-4 Calibrations, across all Abdomen insertion site participants and all days. MARD is calculated by absolute value of [(sensor glucose value - YSI glucose value) / YSI glucose value] * 100
Time Frame: Days 1, 3 and 6 of sensor wear
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- All Subjects With Abdomen Insertion: This group contains all subjects with sensors inserted in the abdomen
Arm/Group | All Subjects With Abdomen Insertion
Number analyzed (Participants) | 61
percentage of difference | 13.6 (13.6)

4. Other Pre Specified Outcome: Mean Absolute Relative Difference (MARD) Between Sensor and YSI for Abdomen Insertion Site, With Calibration Every 12 Hours
Description: This is a measure of Mean Absolute Relative Difference (MARD) between the sensor and the paired YSI plasma glucose value for sensors inserted in the Abdomen insertion site, with Calibration every 12 hours, across all Abdomen insertion site participants and all days. MARD is calculated by absolute value of [(sensor glucose value - YSI glucose value) / YSI glucose value] * 100
Time Frame: Days 1, 3 and 6 of sensor wear
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- All Subjects With Abdomen Insertion: All subjects that enrolled in the study and had sensors inserted in the abdomen insertion area.
Arm/Group | All Subjects With Abdomen Insertion
Number analyzed (Participants) | 61
percentage of difference | 14.7 (13.7)

5. Other Pre Specified Outcome: Mean Absolute Relative Difference (MARD) Between Sensor and YSI for Buttock Insertion Site, With 3-4 Calibrations Throughout the Day
Description: This measure is the Mean Absolute Relative Difference (MARD) between sensor glucose value and paired YSI plasma glucose measurement for sensors inserted in the Buttock insertion site, with 3-4 Calibrations, across all Buttock insertion site participants and all days. MARD is calculated by absolute value of [(sensor glucose value - YSI glucose value) / YSI glucose value] * 100
Time Frame: Days 1, 3 and 6 of sensor wear
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- All Subjects With Buttock Insertion: All subjects that enrolled in the study who had sensors inserted in the buttock insertion site.
Arm/Group | All Subjects With Buttock Insertion
Number analyzed (Participants) | 61
percentage of difference | 15.5 (16.0)

6. Other Pre Specified Outcome: Mean Absolute Relative Difference (MARD) Between Sensor and YSI for Buttock Insertion Site, With Calibration Every 12 Hours
Description: This measure is the Mean Absolute Relative Difference (MARD) between sensor glucose values and paired YSI plasma glucose values for sensors inserted in the Buttock insertion site, with Calibration every 12 hours, across all Buttock insertion site participants and all days. MARD is calculated by absolute value of [(sensor glucose value - YSI glucose value) / YSI glucose value] * 100
Time Frame: Days 1, 3 and 6 of sensor wear
Measure: Mean (Standard Deviation); unit: percentage of difference
Groups:
- All Subjects With Buttock Insertion: All subjects who enrolled in the study and had sensors inserted in the buttock insertion area.
Arm/Group | All Subjects With Buttock Insertion
Number analyzed (Participants) | 61
percentage of difference | 18.2 (23.8)

ADVERSE EVENTS:
Time Frame: Severe adverse event data and adverse event data were collected during the 2-4 weeks study duration
Groups:
- All Completed Subjects: All subjects that completed the study
Arm/Group | All Completed Subjects
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 17/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Completed Subjects (N=90)
Nausea (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Chest Pain (General disorders) | 1 (1)
Application Site Pain (General disorders) | 1 (1)
Edema L Hand (General disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 3 (3)
Flu (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Skin Infection (Infections and infestations) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Pain in Arm (Musculoskeletal and connective tissue disorders) | 2 (4)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arm Discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Sinus Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less